CLINICAL TRIAL: NCT00926393
Title: A Phase IV, Multi-center, Double-blind, Double-dummy, Randomized, Parallel-group Study to Compare the Tolerability of Quetiapine Fumarate Immediate Release (Seroquel IR) With Quetiapine Fumarate Extended Release (Seroquel XR) During Initial Dose Escalation in Patients With Bipolar Depression
Brief Title: Study Comparing the Tolerability of Seroquel IR With Seroquel XR in Patients With Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans Eriksson, MD, Medical Science Sr Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: D1443C00040
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Results first posted 2011-03-31 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Bipolar Depression
Keywords: inpatient; bipolar depression; quetiapine; Seroquel IR; Seroquel XR; safety; tolerability
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine Immediate Release (IR) (Active Comparator): Quetiapine 25, 100, 200 and 300 mg
  Interventions: Drug: Quetiapine Immediate Release
- Quetiapine Extended Release (XR) (Active Comparator): Quetiapine 50, 200, 300
  Interventions: Drug: Quetiapine Extended Release

INTERVENTIONS:
Drug: Quetiapine Immediate Release — Oral, 3 tablets daily: (2 x 25 mg + 1 x 50 mg) at one time each day
  Other Names: Seroquel IR
  Arms: Quetiapine Immediate Release (IR)
Drug: Quetiapine Extended Release — Oral, 3 tablets daily: (2 x 25 mg + 1 x 50 mg) at one time each day
  Other Names: Seroquel XR
  Arms: Quetiapine Extended Release (XR)

SUMMARY:
The purpose of the study is to compare the sedation profile one hour after dose administration between Seroquel IR and Seroquel XR.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR documented bipolar I or bipolar II, most recent episode depressed
* Outpatient status as enrollment

Exclusion Criteria:

* Other than bipolar disorder under study, patients must not have another current, major disorder that is symptomatic or has required treatment within 6 months of enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Datto, MD, Study Director — AstraZeneca

REFERENCES:
- [Derived] Riesenberg RA, Baldytcheva I, Datto C. Self-reported sedation profile of quetiapine extended-release and quetiapine immediate-release during 6-day initial dose escalation in bipolar depression: a multicenter, randomized, double-blind, phase IV study. Clin Ther. 2012 Nov;34(11):2202-11. doi: 10.1016/j.clinthera.2012.09.002. Epub 2012 Oct 8. PMID 23059166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A 7-day, inpatient, multicenter, double-blind, double-dummy, randomized, parallel group, Phase IV study was done to compare the tolerability of quetiapine IR with quetiapine XR during initial dose escalation in patients with bipolar depression. In total 139 patients were randomized in 15 centers in the USA between June and August 2009.
Pre-assignment Details: Patients must have DSM-IV-TR documented bipolar I or bipolar II, most recent episode depressed, and outpatient status at enrollment . Patients must not have another current, major disorder that is symptomatic or has required treatment within 6 months of enrollment.
Groups:
- Quetiapine IR: Quetiapine fumarate Immediate Release
- Quetiapine XR: Quetiapine fumarate Extended Release
Period: Overall Study
Arm/Group | Quetiapine IR | Quetiapine XR
Started | 69 | 70
Completed | 67 | 67
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine IR | Quetiapine XR | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Customized [Number; unit: Participants]
  18-39 | 28 | 31 | 59
  40-50 | 41 | 39 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 66
  Male | 37 | 36 | 73

OUTCOME MEASURES:

1. Primary Outcome: Modified Bond-Lader Visual Analog Scale Score After 50-mg Dose (Day 2)
Description: The Modified Bond-Lader Visual Analog Scale (VAS) uses a 100 mm line, each with a set of opposing adjectives at either end:Alert (=0) - Drowsy (=100); If patient is sleeping the Bond-Lader VAS will be assign a score of 100.
Time Frame: At 1 hour post-dose, Day 2 (50 mg)
Population: The modified intent-to-treat (MITT) analysis data set included all randomized patients who received study treatment, classified according to their randomized treatment and provided the Modified Bond-Lader VAS score at baseline (pre-dose at Day 1 or Day 2) and at least 1 hour after 50 mg dose administration.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 65 | 69
units on scale | 45.022 [38.287 to 51.758] | 32.472 [25.935 to 39.009]

2. Secondary Outcome: Modified Bond-Lader Visual Analog Scale Score After 100-mg Dose (Day 3)
Description: as for outcome 1
Time Frame: At 1 hour post-dose, Day 3 (100 mg)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 65 | 69
units on scale | 51.521 (3.341) [lower limit 3.341] | 29.146 (3.239) [lower limit 3.239]

3. Secondary Outcome: Modified Bond-Lader Visual Analog Scale Score After 200-mg Dose (Day 4)
Description: as for outcome 1
Time Frame: At 1 hour post-dose, Day 4 (200 mg)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 65 | 69
units on scale | 48.336 (3.703) [lower limit 3.703] | 30.130 (3.609) [lower limit 3.609]

4. Secondary Outcome: Modified Bond-Lader Visual Analog Scale Score After 300-mg Dose (Day 5)
Description: as for outcome 1
Time Frame: At 1 hour post-dose, Day 5 (300 mg)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 65 | 69
units on scale | 49.414 (4.347) [lower limit 4.347] | 32.626 (4.258) [lower limit 4.258]

5. Secondary Outcome: Modified Bond-Lader Visual Analog Scale Score After 300-mg Dose (Day 6)
Description: as for outcome 1
Time Frame: At 1 hour post-dose, Day 6 (300 mg)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 65 | 69
units on scale | 48.959 (4.015) [lower limit 4.015] | 30.144 (3.910) [lower limit 3.910]

6. Secondary Outcome: Maximum Intensity Modified Bond-Lader Visual Analog Scale Score
Description: The Maximum Intensity Modified Bond-Lader VAS after dose (MaxIntVAS) is calculated as maximum possible value of VAS during that day at any from 1, 2, 3, 4, 5, 12, 13, 14 hours post-dose assessments
Time Frame: During Day 2 (50 mg)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 65 | 69
units on scale | 99.929 (1.353) [lower limit 1.353] | 96.937 (1.313) [lower limit 1.313]

7. Secondary Outcome: Time to Maximum Intensity Modified Bond-Lader Visual Analog Scale Score
Description: Time (Tmax) to Maximum Intensity Modified Bond-Lader VAS after dose is corresponding assessment time (one from 1, 2, 3, 4, 5, 12, 13, 14 hours post-dose) of MaxIntVas
Time Frame: During Day 2 (50 mg)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 65 | 69
Hours | 3.685 (0.246) [lower limit 0.246] | 4.254 (0.239) [lower limit 0.239]

8. Secondary Outcome: Area Under the Modified Bond-Lader Visual Analog Scale-time Curve
Description: Area under the Modified Bond-Lader VAS-time curve is calculated by the linear trapezoidal formula which equals sum of (Ck+Ck+1)/2 multiplied by the time interval between k and k+1 observations, where Ck and Ck+1 are the corresponding the intensity of sedation evaluations measured by the Modified Bond-Lader VAS from 1 to 14 hours post-dose
Time Frame: During Day 2 (50 mg)
Population: The randomized safety analysis data set included all patients who received at 1 dose of randomized study treatment during the Randomized treatment Phase, classified according to actual treatment taken.
Measure: Least Squares Mean (Standard Error); unit: mm * hour
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 65 | 69
mm * hour | 1061.12 (31.559) [lower limit 31.559] | 988.842 (30.612) [lower limit 30.612]

9. Secondary Outcome: Change in Simpson-Angus Scale (SAS) Total Score
Description: SAS total score is the sum of the 10 individual-item scores (range:0-40), with the score for each item ranging from 0 to 4, higher scores indicate greater severity of Parkinsonian symptoms. Change : total score at day 7 minus total score at randomization. Increase in Change of total score indicates an increase in extrapyramidal motor symptoms.
Time Frame: Randomization to Day 7
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 69 | 70
units on scale | -0.1 (0.8) | 0.1 (0.5)

10. Secondary Outcome: Change in Barnes Akathisia Rating Scale (BARS) Global Score
Description: BARS global score is the 4th individual-item score on the BARS scale,the Global Assessment of Akathisia, with the score ranging from 0 to 5. Change : score at day 7 minus score at randomization. Increase in Change of BARS global score indicates an increase in akathisia.
Time Frame: Randomization to Day 7
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 69 | 70
units on scale | -0.07 (0.43) | -0.09 (0.45)

11. Secondary Outcome: Change in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: AIMS total score is the sum of the 10 individual-item scores (range:0-40), with the score for each item ranging from 0 to 4. Change : total score at day 7 minus total score at randomization. Increase in Change of total score indicates an increase in abnormal voluntary movements.
Time Frame: Randomization to Day 7
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 69 | 70
units on scale | -0.01 (0.3) | -0.04 (0.4)

12. Secondary Outcome: Number of Patients With Potential Extrapyramidal Symptoms (EPS)
Description: Number of patients with adverse events potentially associated with EPS collected by MedDRA Preferred Terms as akathisia, extrapyramidal disorder, restlessness
Time Frame: From start of the study treatment to last dose plus 30 days
Population: as for outcome 8
Measure: Number; unit: Patients
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 69 | 70
Patients | 8 | 2

13. Secondary Outcome: Number of Patients With Potential Somnolence
Description: Number of patients with adverse events potentially associated with somnolence collected by MedDRA Preferred Terms as lethargy, sedation, somnolence
Time Frame: From start of the study treatment to last dose plus 30 days
Measure: Number; unit: Patients
Arm/Group | Quetiapine IR | Quetiapine XR
Number analyzed (Participants) | 69 | 70
Patients | 11 | 12

ADVERSE EVENTS:
Arm/Group | Quetiapine IR | Quetiapine XR
Serious Adverse Events (participants affected / at risk) | 0/69 | 3/70
Other Adverse Events (participants affected / at risk) | 33/69 | 29/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine IR (N=69) | Quetiapine XR (N=70)
Convulsion (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine IR (N=69) | Quetiapine XR (N=70)
Dry Mouth (Gastrointestinal disorders) | 9 | 15
Increased Appetite (Metabolism and nutrition disorders) | 11 | 11
Dizziness (Nervous system disorders) | 11 | 4
Headache (Nervous system disorders) | 8 | 4
Somnolence (Nervous system disorders) | 5 | 7
Fatigue (General disorders) | 3 | 6
Sedation (Nervous system disorders) | 4 | 5
Tachycardia (Cardiac disorders) | 6 | 3
Akathisia (Nervous system disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to collaborate in good faith with AstraZeneca with regards to the contents and formation of any publication or disclosure to be made by the PI and to pay due consideration to the comments, views and opinions offered by AstraZeneca